CLINICAL TRIAL: NCT06783452
Title: Investigation of the Effectiveness of Clinical Pilates in Hip Osteoarthritis: A Randomised Controlled Trial
Brief Title: Clinical Pilates in Hip Osteoarthritis: A Randomised Controlled Trial
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Sevtap Günay, associate professor, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KatipCelebiUniversityIzmır
Record Dates: First submitted 2025-01-07; First posted 2025-01-20 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Hip Osteoarthritis
Keywords: pilates; exercise; pain; osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip; Motor Activity; Pain; Osteoarthritis | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clinical Pilates Group (Experimental): The patients participated in a Clinical Pilates program under the supervision of a physiotherapist twice a week for a duration of 12 weeks.
  Interventions: Other: Exercise
- Conventional Therapeutic Exercise Program (Experimental): The patients participated in a Conventional Therapeutic Exercise program under the supervision of a physiotherapist twice a week for a duration of 12 weeks.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Clinical Pilates Session:
  Each clinical Pilates movement will have three difficulty levels: beginner, intermediate, and advanced. The progression criteria for increasing difficulty will be determined by the prevention of compensatory movements, the ability to activate target muscles, achieving more controlled movements during exercise, and maintaining a more stable posture. This program will include standard hip-focused as well as full-body clinical Pilates movements.
  Arms: Clinical Pilates Group
Other: Exercise — Conventional Therapeutic Exercise Program:
  The Conventional Therapeutic Physiotherapy Exercise Program will consist of strengthening exercises for the hip flexors, extensors, abductors, and adductors, as well as the knee flexors and extensors. Additionally, stretching exercises for the hip flexors, extensors, abductors, and adductors, as well as the knee flexors and extensors, will be included. Stretching exercises will be performed at a pain-free point where tension is felt, holding for 10-30 seconds to achieve a total duration of 60 seconds per muscle group. These exercises will represent standard hip-targeted exercises.
  During the exercises, patients will be asked to rate their perceived exertion using the BORG scale (0-10). When the difficulty level reaches 5-6 points, progression will first be achieved by increasing the number of sets, followed by the use of resistance bands.
  Arms: Conventional Therapeutic Exercise Program

SUMMARY:
The aim of this study is to investigate the effect of a clinical Pilates exercise program on reducing symptoms in individuals with hip osteoarthritis. The main questions it aims to answer are:

* Does a clinical Pilates exercise program have an effect on pain, range of motion, physical function, performance, spinal mobility, postural control, disability, self-efficacy, and quality of life in individuals with hip osteoarthritis?
* Does a conventional therapeutic exercise program have an effect on pain, range of motion, physical function, performance, spinal mobility, postural control, disability, self-efficacy, and quality of life in individuals with hip osteoarthritis? Researchers will compare clinical pilates program to conventional therapeutic exercise program to see if exercise works to reducing hip osteoarthritis symptoms.

Participants will:

* Take clinical pilates or Conventional Therapeutic Exercise twice a week for 12 weeks
* The patients will be assessed by a blind evaluator both before and after the treatment.

DETAILED DESCRIPTION:
The clinical Pilates group will perform 45-minute exercise sessions under the supervision of a physiotherapist twice a week for 12 weeks, focusing on fundamental spinal alignments and Pilates principles. The program will include exercises that engage all body segments and combine movement with breathing. Participants will progress to more advanced levels as long as they can maintain proper alignment. Clinical Pilates exercises are structured into three levels of difficulty, and participants who complete the current level without compromising alignment will advance to the next level. The Conventional Therapeutic Exercise group will participate in an exercise program under the supervision of a physiotherapist twice a week for 12 weeks. The program, consisting of stretching and strengthening exercises, will last approximately 45 minutes. Resistance bands will be used to facilitate progression. Based on the individual's perceived difficulty level, resistance bands will be introduced or adjusted by changing their color to increase or decrease resistance.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Diagnosis of hip osteoarthritis (OA) according to the American College of Rheumatology
* Not on the waiting list for hip replacement surgery
* Willingness to participate in the exercise program

Exclusion Criteria:

* Symptomatic OA in the knee or big toe
* Presence of other types of arthritis
* History of hip and/or knee prosthesis or fracture
* Use of walking aids
* Regular exercise habit of two or more sessions per week
* Corticosteroid injection into the hip within the past 12 months
* Participation in a physical therapy program for hip pain within the past 3 months
* Severe cardiovascular disorders or other comorbidities that significantly limit daily physical capacity or contraindicate physical exertion

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-11-30 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | From enrollment to the end of treatment at 12 weeks
  Pain intensity will be evaluated using the Visual Analog Scale (VAS). During the assessment, patients will be asked to mark the degree of pain they feel on a 100-mm horizontal line. The distance from the starting point to the marked point will be measured with a ruler, and the pain intensity will be recorded in millimeters.
  The VAS, developed by Vas Price et al. (1983), is a validated and reliable tool for determining the perceived intensity of pain. It is simple to administer and widely used in clinical practice.
Lumbopelvic Stabilization | From enrollment to the end of treatment at 12 weeks
  Lumbopelvic stabilization will be assessed using the "Stabilizer Pressure Biofeedback Unit". Prior to the measurement, each participant will be instructed in the corset technique for contracting the Transversus Abdominis muscle while lying in a supine position. Participants will be asked to lie on their back with their knees bent (hook-lying position), maintaining a neutral and relaxed spinal alignment.
  A pressure cell, inflated with air and connected to a stabilizer, will be placed under the lumbar spine. The manometer's baseline pressure will be inflated to 40 mmHg. Participants will then be instructed to contract their Transversus Abdominis muscle using the abdominal corset technique without moving the spine or pelvis and without holding their breath. They will be required to maintain this contraction for 5 seconds.
  After three practice trials to ensure learning, participants will rest for 30 seconds. The actual measurement will consist of three repetitions of 10 seconds each.

SECONDARY OUTCOMES:
Postural Control: | From enrollment to the end of treatment at 12 weeks
  Static balance assessment was performed using a proprioceptive-stabilometric assessment machine (ProKin 252; TecnoBody, Prokin, Italy). The device consists of a force platform with a 55 cm diameter surface, a sampling rate of 20 Hz, and a sensitivity of 0.1.
  For all participants, anterior-posterior stability, medial-lateral stability index, and total stability index were measured under two conditions: with eyes open and eyes closed. Participants were instructed to stand motionless on the fixed platform surface for 30 seconds with their eyes open. During this time, the minimal postural sway of the body was recorded by the device, and a report was generated. The same measurement was then repeated with eyes closed.
  Higher scores indicate impaired postural stability, while lower scores represent normal postural stability
The Active Normal Range of Motion | From enrollment to the end of treatment at 12 weeks
  The Active Normal Range of Motion (ANROM) of the participants will be evaluated in appropriate positions. If necessary, measurements will be taken using a universal goniometer, and the degree of limitation will be recorded.
  In the supine position, hip flexion, abduction, and adduction ANROM will be assessed, while hip extension ANROM will be evaluated in the prone position.
Physical Function | From enrollment to the end of treatment at 12 weeks
  The physical function levels of the participants will be measured using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). This assessment tool consists of three subscales: Section A evaluates pain severity, Section B assesses joint stiffness, and Section C measures physical function.
  The scale includes 5 questions for pain, 2 questions for joint stiffness, and 17 questions for physical function. Each question is scored on a scale from 1 to 5, where:
  1. = None
  2. = Mild
  3. = Moderate
  4. = Severe
  5. = Very Severe
  Each subscale generates a total score independently. A lower score indicates better health status, while a higher score reflects worse health status. The scoring ranges are as follows:
  Section A (pain): 5-25 Section B (joint stiffness): 2-10 Section C (physical function): 17-85
Disability | From enrollment to the end of treatment at 12 weeks
  The disability levels of participants will be assessed using the Hip Disability and Osteoarthritis Outcome Score-Physical Function Short Form (HOOS-PS). HOOS-PS is a 5-item scale designed to evaluate symptoms and functional status related to hip osteoarthritis. This questionnaire was developed by OMERACT/OARSI.
  Each question is scored on a scale of 0 to 4 based on the degree of difficulty, with a maximum possible score of 20. However, the scores are normalized to a range of 0-100, where 0 indicates the best functional status.
Self-Efficacy | From enrollment to the end of treatment at 12 weeks
  The self-efficacy levels of participants will be assessed using the Arthritis Self-Efficacy Scale. This scale consists of 20 items evaluated on a 10-point visual scale and includes three subdimensions: self-efficacy for pain, self-efficacy for function, and self-efficacy for other symptoms.
  Self-efficacy for pain involves the perception of the ability to reduce pain and maintain it at a low level. The first 5 items of the scale belong to this subdimension.
  Self-efficacy for function measures the ability to perform functions affected by arthritis, particularly in the hand and foot joints. The next 9 items following the first 5 are included in this subdimension.
  Self-efficacy for other symptoms evaluates the ability of individuals with arthritis to cope with existing symptoms. The final 6 items fall under this subdimension.
  Each item is scored on a 10-point scale, ranging from "Not at all confident = 1" to "Very confident = 10." The total score can range from 20 (minimu
Quality of Life Index | From enrollment to the end of treatment at 12 weeks
  The quality of life levels of the participants will be evaluated with SF-12. SF-12 consists of 8 sub-dimensions and 12 items including physical functioning (2 items), physical role (2 items), body pain (1 item), general health (1 item), energy (1 item), social functioning (1 item), emotional role (2 items) and mental health (2 items). The items related to physical and emotional role are answered as 'yes or no', while the other items have Likert-type options ranging between 3 and 6. Physical component summary (PCS)-12 score is obtained from general health, physical functioning, physical role and body pain sub-dimensions, while mental component summary (MCS)-12 score is obtained from social functioning, emotional role, mental health and energy sub-dimensions. Both FCI-12 and MCI-12 scores ranged from 0 to 100, with higher scores representing better health.
30-Second Chair Stand Test | From enrollment to the end of treatment at 12 weeks
  The participant is asked to sit upright on a standard 43 cm high chair with their arms crossed over their shoulders. They are then instructed to stand up and sit down as many times as possible in 30 seconds, at the fastest pace they can. They are told that they can rest if they get tired. The number of stand-ups is recorded.
40-Meter Fast Walk Test | From enrollment to the end of treatment at 12 weeks
  The participant is asked to walk as fast as they can, but not run, for a distance of 40 meters. The time taken to complete the test is recorded.
Stair Climbing Test | From enrollment to the end of treatment at 12 weeks
  The participant is asked to climb up a 9-step stair, turn around, and climb back down. The time taken is recorded, and their ability to perform the functional task is observed.
Timed Up and Go Test | From enrollment to the end of treatment at 12 weeks
  The participant is asked to stand up from a chair, walk 3 meters, turn around, walk back to the chair, and sit down. The time taken to complete the test is recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk Training and Research Hospital, Izmir, Turkey (Türkiye)

REFERENCES:
- [Background] Rego TAM, Ferreira APL, Villela DW, Shirahige L, Xavier AB, Braz RRS, Guerino MR, Araujo MDGR. Effects of mat Pilates on older adult women with knee osteoarthritis: A randomized controlled trial. J Bodyw Mov Ther. 2023 Jan;33:136-141. doi: 10.1016/j.jbmt.2022.02.007. Epub 2022 Apr 15. PMID 36775508
- [Background] Patti A, Zangla D, Sahin FN, Cataldi S, Lavanco G, Palma A, Fischietti F. Physical exercise and prevention of falls. Effects of a Pilates training method compared with a general physical activity program: A randomized controlled trial. Medicine (Baltimore). 2021 Apr 2;100(13):e25289. doi: 10.1097/MD.0000000000025289. PMID 33787615
- [Background] Gebhart JJ, Weinberg DS, Bohl MS, Liu RW. Relationship between pelvic incidence and osteoarthritis of the hip. Bone Joint Res. 2016 Feb;5(2):66-72. doi: 10.1302/2046-3758.52.2000552. PMID 26912384
- [Background] Bannuru RR, Osani MC, Vaysbrot EE, Arden NK, Bennell K, Bierma-Zeinstra SMA, Kraus VB, Lohmander LS, Abbott JH, Bhandari M, Blanco FJ, Espinosa R, Haugen IK, Lin J, Mandl LA, Moilanen E, Nakamura N, Snyder-Mackler L, Trojian T, Underwood M, McAlindon TE. OARSI guidelines for the non-surgical management of knee, hip, and polyarticular osteoarthritis. Osteoarthritis Cartilage. 2019 Nov;27(11):1578-1589. doi: 10.1016/j.joca.2019.06.011. Epub 2019 Jul 3. PMID 31278997